CLINICAL TRIAL: NCT01882621
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial of Monosialoganglioside(GM1) Preventing Neurotoxicity Induced by First-line Chemotherapy Contained Cisplatin in Non-small Cell Lung Cancer Patients.
Brief Title: Monosialoganglioside(GM1) Preventing Neurotoxicity Induced by Cisplatin Contained Chemotherapy in NSCLC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GM1-0324
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Monosialoganglioside(GM1); neurotoxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neurotoxicity Syndromes | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monosialoganglioside(GM1) (Active Comparator): Monosialoganglioside(GM1)80mg + N.S 250ml,qd,D0-D3
  Interventions: Drug: Monosialoganglioside(GM1)
- normal saline (Placebo Comparator): placebo 80mg + N.S 250ml,qd,D0-D3
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Monosialoganglioside(GM1) — 80mg,ivdrip (in the vein) on day 0 - day 3 of each 21 day cycle. Number of Cycles: 4-6 cycles.
  Other Names: Monosialotetrahexosylganglioside Sodium Injection
  Arms: Monosialoganglioside(GM1)
Drug: normal saline — 80mg,ivdrip(in the vein) on day 0-3 of each 21 day cycle. Number of Cycles: 4-6 cycles.
  Arms: normal saline

SUMMARY:
Evaluate the efficacy and safety of Monosialoganglioside(GM1) to prevent the neurotoxicity induced by cisplatin

DETAILED DESCRIPTION:
NSCLC patients received a cisplatin-based doublet chemotherapy are included in this trial. Patients are randomly assigned into the experimental group and control group based on segmented block randomized method. After enrollment, patients should complete four or six chemotherapy and GM1/placebo injection. During the 3w per cycle chemotherapy, cisplatin injection is conducted in D1/D1-3, GM1/placebo (80mg+250ml N.S) is injected from D0 to D3. Neurotoxicity evaluation and quality of life (FACT-NTX and EROTC scale) assessment will be conducted every cycle and 3w/11w/19w after the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytological and histological confirmation of non-small cell lung cancer (NSCLC) diagnosis, single sputum cytology diagnosis is not accepted
* Expected survival period is more than 3 months
* Enough blood function reservation: absolute neutrophil count (ANC) 2 x 10E9/L or higher;platelet count 100 x 109 /L or higher;hemoglobin 9 g/dL or higher.
* Enough liver function reservation:the total bilirubin less than upper limit of normal;AST and ALT acuities were less than 2.5 times the upper limit of normal (ULN);Alkaline phosphatase 5 times the upper limit of normal (ULN) or less.
* Clinical doctors identify patients suitable for standard doses of ganglioside drug therapy, and expected time of medication is at least six weeks
* Within 4 weeks before treatment, did not receive other adverse reaction of drugs may cause similar neurotoxicity; 18 weeks before, did not received platinum-based drugs chemical treatment.
* No more than 1 degree of the peripheral nervous system diseases exists before enrollment, also no other symptom or disease could affect the adverse reactions of neurotoxicity pathological.
* Can't accept other adverse reactions may prevent neurotoxicity treatment or care after enrollment.
* Sign the informed consent form.

Exclusion Criteria:

* Patients with poor general condition, PS score more than 2 points
* Women in pregnancy or lactation
* Patients (male or female) have fertility possibility but not willing to or not to adopt effective contraception
* With other neurological dysfunction which can cause inaccurate record of the occurrence of neurotoxicity and severity
* Known or assignment of any of these products to test drugs allergic agent composition
* Doctors think inappropriate for patients with ganglioside medication or estimated time of less than 6 weeks
* Active infection (determined by the researcher)
* According to the researcher's judgment, there is serious disease to endanger the safety of patients, or may prevent the patients from completing the study
* Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
incidence rate of neurotoxicity adverse events | up to 19 weeks after cisplatin chemotherapy

SECONDARY OUTCOMES:
neurotoxicity adverse events alleviation time | up to 19 weeks after the cisplatin based chemotherapy

OTHER OUTCOMES:
the quality of life of patients | up to 19 weeks after the cisplatin based chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: LI Zhang, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China